CLINICAL TRIAL: NCT03556085
Title: Clinical Evaluation of the Serenity River Stent System to Treat Idiopathic Intracranial Hypertension
Brief Title: Venous Sinus Stenting With the River Stent in IIH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Serenity Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: River 1111-001
Record Dates: First submitted 2018-05-22; First posted 2018-06-14 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: idiopathic intracranial hypertension; venous sinus stenting
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single arm, open label clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Venous sinus stenting (Experimental): Subjects will have stenting of the transverse-sigmoid sinus
  Interventions: Device: Venous sinus stenting (Serenity River)

INTERVENTIONS:
Device: Venous sinus stenting (Serenity River) — Patient is placed under general anesthesia. From femoral vein access, a standard guide-catheter is advanced in the internal jugular vein (on the side considered for stenting). The sigmoid then transverse sinus is catheterized with a microcatheter and guide-wire and an exchange guide-wire is placed in the superior sagittal sinus. The River stent delivery catheter is advanced over the exchange guide-wire in the sigmoid then transverse sinus up to the torcula. The River stent is deployed to cover the entire transverse sinus and the proximal half of the sigmoid sinus. The catheters are removed and hemostasis obtained by using a closure device or manual compression. The patient is kept overnight in the hospital for observation.

SUMMARY:
The objective of the study is to show that stenting the transverse-sigmoid sinus with the River stent is safe and has probable benefit to relieve clinical symptoms in subjects with idiopathic intracranial hypertension (IIH).

The study will enroll 39 IIH subjects with moderate to severe visual field loss or severe headaches that have failed medical therapy.

The primary safety endpoint is the rate of major adverse event at 12 months The primary probable benefit endpoint is a composite at 12 months of absence of significant sinus stenosis and clinically relevant improvement.

DETAILED DESCRIPTION:
Study objective: The objective of the study is to show that stenting the transverse-sigmoid sinus with the River stent is safe and has probable benefit to relieve clinical symptoms in subjects with idiopathic intracranial hypertension (IIH)

Investigational product: Serenity River Stent System

Study design: prospective, multicenter, single arm, open label clinical trial

Subject population: IIH subjects with significant (>50%) stenosis of the transverse-sigmoid sinuses and moderate to severe visual field loss or severe headaches that have failed medical therapy. In the absence of this trial, subjects would have been offered a surgical treatment of IIH such as sinus stenting with an off-label device, cerebrospinal fluid shunting, or optic nerve sheath fenestration by the treating physician.

* For subjects with visual field loss: if moderate to severe visual field loss (mean deviation between -6db and -30 db) for at least 2 weeks despite escalation of acetazolamide to 1000 mg twice a day or if the visual field deteriorates by more than 2 db during treatment, or treatment intolerance.
* For subjects with headaches: if they have severe headaches (HIT > 59) for at least 4 weeks despite treatment with topiramate 100 mg twice a day or other headache medication, or treatment intolerance.

Enrollment size and sites: 39 subjects will be enrolled in up to 10 US sites.

Primary safety endpoint: Major Adverse Event at 12 months. The MAE is a composite of the following: moderate or severe stroke (NIHSS > 3), neurological death, perforation or thrombosis of sinus or cerebral vein, device distal embolization, need for target lesion revascularization or need for alternate IIH surgical procedure such as cerebrospinal fluid shunting or optic nerve sheath fenestration.

Primary probable benefit endpoint: a composite at 12 months of:

* Absence of significant (>50%) stenosis of the stented sinus on retrograde catheter venography and
* Trans-stent pressure gradient < 8 mm Hg and
* Clinically relevant improvement in the main clinical outcome per specific inclusion criteria and stabilization or better of the other:

  * Headaches: if the specific inclusion criteria was headaches, improvement in the HIT- 6 scale by > 4 points and improvement or stabilization of visual field.
  * Ophthalmic: if the specific inclusion criteria was visual field loss, improvement of visual field by > 29% of the baseline value in the study eye, stabilization or improvement in the fellow eye, and improvement or stabilization of headaches.

Study duration and follow-up: The subjects will be followed at 2 weeks, 3 months, 6 months and 12 months. At 12 months, clinical examination, lumbar puncture and retrograde catheter venography with manometry will be performed to evaluate the patency of the treated sinus and the absence of trans-stent pressure gradient. Subjects will be consented to be clinically followed annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for participation in the study:

1. Subject is > 18 year-old and has given informed consent.
2. Diagnosis of IIH per Modified Dandy Criteria.
3. CSF opening pressure is > 25 cm H2O.
4. Radiological examination (magnetic resonance venography (MRV) or computed tomographic venography (CTV)) shows bilateral transverse-sigmoid venous sinus stenosis (> 50%) or unilateral stenosis of the dominant sinus with contralateral hypoplastic sinus.
5. Presence of IIH clinical symptoms (6. OR 7.)
6. Headaches: Score > 59 (severe impact) on the HIT-6 scale, refractory to medical therapy (e.g. acetazolamide 1000 mg twice daily, topiramate 100 mg twice daily, or other headache medication) for ≥ 4 weeks, or treatment intolerance OR
7. Visual field loss: defined by perimetric mean deviation (PMD) between -6 dB and -30 dB in one or both eyes (with papilledema Grade >1) despite at least 2 weeks of medical therapy with acetazolamide 1000 mg twice daily, or if the visual field deteriorates by more than 2 dB during treatment, or treatment intolerance.
8. In the absence of this study, the subject would have been offered a surgical intervention by Optic Nerve Sheath Fenestration (ONSF), Cerebro Spinal Fluid (CSF) shunting procedure, or venous sinus stenting with an off-label device.
9. Catheter manometry shows a pressure gradient > 8 mm Hg across the transverse sigmoid sinus stenosis.
10. Venographic evidence of sinus stenosis (> 50%)

Exclusion Criteria:

Subject must be excluded from participation in this study if any of the following criteria are met

1. Subjects presenting with de novo papilledema and severe visual field(VF) deficit (VF loss > -15db) that requires immediate surgical treatment without prior attempt of medical therapy.
2. Currently has or plans to have an implanted CSF shunt.
3. History of previously implanted intra-cranial sinus stent.
4. Transverse-sigmoid sinus vessel size <5 mm or >10 mm.
5. Creatinine > 1.5 mg/dl and/or creatinine clearance < 60 mL/min (except if patients is already on hemodialysis).
6. Allergic to imaging contrast media (iodine or gadolinium) despite premedication.
7. Allergic to nitinol or nickel.
8. Contra-indication to general anesthesia.
9. Contra-indication to aspirin, clopidogrel or other anticoagulant.
10. Hypercoagulable state (Factor V Leiden, Protein C or S deficiency, Anticardiolipin antibodies, Lupus anticoagulant, B2-glycoprotein-1 antibodies, or Hyperhomocysteinemia).
11. Currently requiring full anti-coagulation for other medical reasons, such as atrial fibrillation (AF), artificial valves, deep vein thrombosis pulmonary embolism, etc.
12. History of stroke or transient ischemic attack (TIA).
13. History of AF or other risks of stroke.
14. History of deep vein thrombosis or pulmonary embolism.
15. History of severe chronic obstructive pulmonary disease or other severe respiratory disease.
16. History of severe carotid atherosclerotic disease.
17. History of heart failure, dilated cardiomyopathy, or congenital heart conditions, etc. that are at high thrombogenic risk.
18. History of uncontrolled diabetes.
19. Use (oral) of tetracycline derivative, retinoid or vitamin A during the last 3 months.
20. Cerebral vascular lesions (arteriovenous malformation (AVM), arteriovenous fistula, aneurysms, significant stenosis of extra- or intra-cranial vessels other than the targeted venous sinus stenosis,intracranial artery dissection, etc.).
21. Patient has visions loss due to other disease (e.g. cataract, macular degeneration, glaucoma, etc.).
22. Inability to provide reliable and reproducible visual field examinations (>15% false positive errors and/or failure to maintain fixation for eye monitoring).
23. For female subject of child bearing potential, pregnant or not willing to use contraception for 12 months.
24. Presence of a physical, mental or social condition that could prevent adequate one-year follow-up (homelessness, drug dependency, anticipation of moving far away, life threatening disease, terminal illness).
25. Anatomical anomaly of the venous sinus which would prevent safe catheterization and stenting (e.g multi-channel sinus)
26. Currently enrolled in a premarket investigational study. Enrollment in a post market study that does not impact the River™ Stent procedure or device is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Event (MAE) | 12 months
  The MAE is a composite of the following:
  Moderate or severe stroke (NIH stroke scale > 3) Neurological death Perforation of sinus or cerebral vein Thrombosis of sinus or cerebral vein Device distal embolization Need for target lesion revascularization or need for IIH alternate procedure (cerebrospinal fluid shunting or optic nerve sheath fenestration)
Clinical improvement with no restenosis of the venous sinus | 12 months
  The primary probable benefit endpoint is a composite of:
  1. Absence of significant stenosis (defined as >50% stenosis of reference vessel diameter) of the main dural venous sinus on retrograde catheter venography (RCV) AND
  2. Trans-stent pressure gradient (measured during the RCV) < 8 mm Hg AND
  3. Clinically relevant improvement in the main clinical outcome per specific inclusion criteria (headache or ophthalmic) and stabilization or better of the other

SECONDARY OUTCOMES:
Individual components of MAE. | 12 months
  Components of MAE will be reported as individual event rates.
Cerebrospinal fluid (CSF) opening pressure at 12 months | 12 months
  CSF opening pressure will be measured via lumbar puncture in the lateral decubitus position.
Stent patency at 12 months | 12 months
  Stent patency will be assessed by retrograde catheter venography. Patency is defined as absence of significant (>50%) stenosis
Medications | 12 months
  Change in IIH medications and dosage at 12 months compared to baseline
Headaches | 12 months
  Change in headaches assessed using the Headache Impact Test (HIT-6) scale (minimum score 36, maximum 78; higher value represents worse headache) at 12 months compared to baseline.
Papilledema | 12 months
  Change in papilledema grading using Frisen scale (Stage 0 to 5; stage 0 represents no papilledema and is the best outcome) at 12 months compared to baseline.
Visual acuity | 12 months
  Change in visual acuity using the Early treatment Diabetic Retinopathy (ETDRS) chart at 12 months compared to baseline.
Retinal Nerve Fiber Layer Thickness | 12 months
  Change in retinal nerve fiber layer thickness measured using Optical Coherence Tomography (OCT) at 12 months compared to baseline.
Tinnitus | 12 months
  Change in the intensity of tinnitus evaluated on the Tinnitus Functional Index (TFI) score (overall score; minimum 0, maximum 100; 100 is the worst tinnitus with the worst negative impact) at 12 months compared to baseline.
Quality of Life SF-12 | 12 months
  Change in quality of life assessed with the Short Form health survey 12 items (SF-12) at 12 months compared to baseline
Quality of Life NEI-VFQ-25 | 12 months
  Change in quality of life assessed with the National Eye Institute - Visual Functioning Questionnaire - 25 at 12 months compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Athos Patsalides, MD, Principal Investigator — Northwell Health
Locations (6):
- United States (6):
  - Baptist Health, Jacksonville, Florida
  - UB Neurosurgery, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - Weill Cornell Medicine, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albuquerque FC, Gross BA, Levitt MR. Time to re-assess the treatment of idiopathic intracranial hypertension. J Neurointerv Surg. 2016 Jun;8(6):549-50. doi: 10.1136/neurintsurg-2016-012460. No abstract available. PMID 27178402
- [Result] Abubaker K, Ali Z, Raza K, Bolger C, Rawluk D, O'Brien D. Idiopathic intracranial hypertension: lumboperitoneal shunts versus ventriculoperitoneal shunts--case series and literature review. Br J Neurosurg. 2011 Feb;25(1):94-9. doi: 10.3109/02688697.2010.544781. PMID 21323404
- [Result] Aguilar-Perez M, Martinez-Moreno R, Kurre W, Wendl C, Bazner H, Ganslandt O, Unsold R, Henkes H. Endovascular treatment of idiopathic intracranial hypertension: retrospective analysis of immediate and long-term results in 51 patients. Neuroradiology. 2017 Mar;59(3):277-287. doi: 10.1007/s00234-017-1783-5. Epub 2017 Mar 2. PMID 28255904
- [Result] Ahmed RM, Wilkinson M, Parker GD, Thurtell MJ, Macdonald J, McCluskey PJ, Allan R, Dunne V, Hanlon M, Owler BK, Halmagyi GM. Transverse sinus stenting for idiopathic intracranial hypertension: a review of 52 patients and of model predictions. AJNR Am J Neuroradiol. 2011 Sep;32(8):1408-14. doi: 10.3174/ajnr.A2575. Epub 2011 Jul 28. PMID 21799038
- [Result] Dinkin MJ, Patsalides A. Venous Sinus Stenting in Idiopathic Intracranial Hypertension: Results of a Prospective Trial. J Neuroophthalmol. 2017 Jun;37(2):113-121. doi: 10.1097/WNO.0000000000000426. PMID 27556959
- [Result] Kanagalingam S, Subramanian PS. Cerebral venous sinus stenting for pseudotumor cerebri: A review. Saudi J Ophthalmol. 2015 Jan-Mar;29(1):3-8. doi: 10.1016/j.sjopt.2014.09.007. Epub 2014 Sep 27. PMID 25859134
- [Result] Dinkin MJ, Patsalides A. Venous Sinus Stenting for Idiopathic Intracranial Hypertension: Where Are We Now? Neurol Clin. 2017 Feb;35(1):59-81. doi: 10.1016/j.ncl.2016.08.006. PMID 27886896